CLINICAL TRIAL: NCT00021359
Title: A Phase II Trial of Dexamethasone and 13-cis-Retinoic Acid as First-Line Treatment for Multiple Myeloma
Brief Title: Isotretinoin Plus Dexamethasone in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068772; FCCC-95043 (Other: Fox Chase Cancer Center); NCI-G01-1985 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2001-07-11; First posted 2004-03-11 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Isotretinoin

INTERVENTIONS:
Drug: dexamethasone
Drug: isotretinoin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with dexamethasone may be an effective treatment for multiple myeloma.

PURPOSE: Phase II trial to study the effectiveness of combining isotretinoin and dexamethasone in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and duration of response of patients with multiple myeloma treated with dexamethasone and isotretinoin. II. Determine the toxicity of this regimen in these patients. III. Correlate the changes in serum interleukin (IL)-6, IL-6R, and C-reactive and IL-6R expression on plasma cells in the bone marrow with response in patients treated with this regimen.

OUTLINE: Patients receive oral dexamethasone on days 1-4, 9-12, and 17-20 and oral isotretinoin daily. Treatment repeats every 5 weeks for at least 2 courses in the absence of disease progression, insufficient response, or unacceptable toxicity. Patients achieving adequate response continue treatment for 2 courses after achieving a plateau of monoclonal protein, for a minimum of 6 courses total.

PROJECTED ACCRUAL: A total of 18-36 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed multiple myeloma Elevated monoclonal protein in serum and/or urine

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3* Platelet count at least 75,000/mm3* *Unless secondary to multiple myeloma involvement of the bone marrow Hepatic: Bilirubin less than 1.5 mg/dL Transaminase less than 2 times normal Renal: Creatinine less than 2.0 mg/dL No overt renal insufficiency Cardiovascular: No congestive heart failure No myocardial infarction within the past 6 months No significant arrhythmia or poorly controlled hypertension Pulmonary: No severe pulmonary disease Other: Triglycerides normal No other severe medical illness No active peptic ulcer disease No brittle insulin-dependent diabetes No severe depression or other psychiatric illness No active infection No history of severe ethanol or drug abuse Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Prior palliative radiotherapy allowed Surgery: At least 3 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 1999-08; Primary Completion 2000-07 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell J. Schilder, MD, Study Chair — Fox Chase Cancer Center
Locations (18):
- United States (18):
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Bon Secours-Holy Family Health System, Altoona, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Conemaugh Memorial Hospital, Johnstown, Pennsylvania
  - Saint Mary Regional Center, Langhorne, Pennsylvania
  - North Penn Hospital, Lansdale, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Southern Chester County Medical Center, West Grove, Pennsylvania